CLINICAL TRIAL: NCT01232764
Title: Pressure Ulcer Multi-disciplinary Teams Via Telemedicine (PUMTT): A Cluster Pragmatic Randomised Controlled Trial in Long Term Care
Brief Title: Pressure Ulcer Multi-disciplinary Teams Via Telemedicine (PUMTT): A Trial in Long Term Care
Acronym: PUMTT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Canadian Patient Safety Institute (Other); Central Community Care Access Center (Unknown)
Responsible Party: Principal Investigator, Anita Stern, Researcher, University of Toronto
Allocation: Randomized | Masking: Single | Purpose: Health Services Research
Other Study IDs: 25048
Record Dates: First submitted 2010-10-29; First posted 2010-11-02 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Pressure Ulcers; Multi-disciplinary Wound Care Teams; Remote Support; Digital Wound Photography
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multi-disciplinary wound care team (Experimental): Stepped wedge study design i.e. start date of exposure is randomized.
  Interventions: Other: Exposure to multi-disciplinary wound care team

INTERVENTIONS:
Other: Exposure to multi-disciplinary wound care team — Phase 1: In Person Support (3 mths)
  Advance Practice Nurses (APNs) affiliated with Enhanced Multi-Disciplinary visit LTC facilities on a weekly basis. The APN may communicate with other members of an EMDT via telephone or online.EMDTs will collectively teach and mentor LTC facility wound care teams throughout the study.
  Phase 2: Remote Support (2-11 mths) In the second phase, EMDTs will support LTC facility staff remotely via telephone and online communication, visiting the facilities on an as needed basis only.
  All PU treatment will be based on RNAO evidence-based guidelines (updated in 2007)contextualized to the LTC setting.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of 'enhanced' multi-disciplinary wound care teams (MDTs) vs. 'usual' care teams in Long Term Care (LTC) facilities in Ontario for the treatment of pressure ulcers. LTC facilities with more than 100 beds that are within a 100 km distance from St. Mikes and have a problem with pressure ulcers will be asked to participate. A total of 10 LTC facilities will be randomly selected (i.e. selected by chance) from those that agree to participate.

The 'enhanced' MDT will be an Advance Practice Nurse(APN) with expertise in wound care who has direct access to the wound care team at St. Mikes. This APN will develop treatment plans in consultation with facility staff, providing targeted pressure ulcer treatment education on an ongoing, case by case basis. Care is supported by telemedicine with the use of digital photography and online communication between members of the care team.

This study is a stepped wedge randomized trial, meaning LTC facilities are assigned to a start date for this study totally by chance. Changes in healing rates, wound related pain, cost, number of new pressure ulcers, and number of wounds healed will be measured before, and after the APN is introduced to facilities. In order to gain more insight into how people felt about this model of care, interviews will be held with individuals and groups of staff at 5 randomly selected facilities before, during, and after the study has been completed.

ELIGIBILITY:
Inclusion Criteria:

* LTC facility must be located within the Toronto Central or Central LHIN geographic boundaries.
* LTC facility must be <100 km from the St. Michael's Hospital wound care team.
* LTC facility must be entering data into MDS.
* LTC facility administrator must consent to participate.
* LTC facility must report a PU prevalence rate >5.5% in the 4th quarter 2009 MDS. [This is the average pressure ulcer prevalence rate for Ontario LTC facilities as reported by the Canadian Institute of Health Information (CIHI) in the 4th quarter 2009.]
* Individual with PU (or Substitute Decision Maker (SDM)) must provide informed consent.

Exclusion Criteria:

* LTC facility <100 beds.
* LTC facility >100 km from the St. Michael's Hospital wound care team
* LTC facility reporting a PU prevalence rate < 5.5% in the 4th quarter 2009 MDS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Rate of reduction in wound surface area (cm2/days) | 6 mths

SECONDARY OUTCOMES:
Percentage of wounds healed | 6 mths

CONTACTS AND LOCATIONS:
Locations (1):
- 12 Long Term Care Facilities, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Stern A, Mitsakakis N, Paulden M, Alibhai S, Wong J, Tomlinson G, Brooker AS, Krahn M, Zwarenstein M. Pressure ulcer multidisciplinary teams via telemedicine: a pragmatic cluster randomized stepped wedge trial in long term care. BMC Health Serv Res. 2014 Feb 24;14:83. doi: 10.1186/1472-6963-14-83. PMID 24559218
- See also: Toronto Health Economic Technology Assessment collaborative — http://www.theta.utoronto.ca